CLINICAL TRIAL: NCT02753478
Title: Safety and Feasibility of Intracoronary Hypothermia in Acute Myocardial Infarction
Acronym: SINTAMI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Luuk Otterspoor, MD, Catharina Ziekenhuis Eindhoven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SINTAMI
Record Dates: First submitted 2016-04-04; First posted 2016-04-28 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Myocardial Infarction
Keywords: hypothermia
MeSH Terms: conditions — Myocardial Infarction; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intracoronary hypothermia group (Experimental): Patients who will receive intracoronary hypothermia before and during percutaneous coronary intervention
  Interventions: Other: intracoronary infusion with saline on 22 and 4°C

INTERVENTIONS:
Other: intracoronary infusion with saline on 22 and 4°C — Routine primary percutaneous intervention will be commenced. Patient will be asked to participate in the study.
  Before reperfusion, saline on room temperature will be infused though the occlusion in the infarct related artery using an over the wire balloon catheter during 10 minutes. The balloon will be inflated to prevent reperfusion in that phase. After 10 minutes the balloon will be deflated allowing reperfusion and infusion with saline on 4°C will be continued for 10 minutes. After this, a coronary stent will be placed.

SUMMARY:
Hypothermia may reduce infarct size in patients with acute myocardial infarction if provided before reperfusion. Human studies using systemic cooling methods failed to show a reduction in infarction size. The use of selective intracoronary hypothermia may overcome the problems of systemic cooling.

The hypothesis of this study is that in patients with acute myocardial infarction, the induction of intracoronary hypothermia is safe and feasible.

DETAILED DESCRIPTION:
In acute myocardial infarction, infarct size is directly related to short and long-term mortality and development of chronic heart failure.Therefore, limiting infarct size is of great worth. Therapies to reduce ischemic injury, by primarily primary percutaneous coronary intervention seem to be exhausted. Consequently, there still remains a need for efforts to develop therapies that target reperfusion injury to obtain additional reduction of infarct size.

Therapeutic hypothermia (32 - 35°C) attenuates reperfusion injury and therefore reduces infarct size in a variety of animal models of acute myocardial infarction (AMI), if provided before reperfusion. In human studies this reduction has not been confirmed so far, probably due to the fact that systemic cooling is slow in reducing temperature and therefore target temperature was not reached in time in a substantial number of patients or not reached at all. Furthermore, systemic cooling has side effects such as severe shivering, volume overload and an enhanced adrenergic state. However, subgroups of patients in all randomized clinical trials with anterior myocardial infarction who reached target temperature before reperfusion did show a reduction in infarct size.

To make therapeutic hypothermia into a valuable treatment for AMI, the method of inducing hypothermia has therefore to be modified. This method should be clinical feasible and quick enough to provide myocardial hypothermia before reperfusion, without prolonging symptom-to-balloon times and without the adverse effects of systemic cooling.

In this study the investigators will evaluate the safety and feasibility of intracoronary hypothermia in 10 patients with acute myocardial infarction.

In study patients, routine primary percutaneous intervention will be commenced. Before reperfusion, saline on room temperature will be infused though the occlusion in the infarct related artery using an over the wire balloon catheter during 10 minutes. The balloon will be inflated to prevent reperfusion in that phase. After 10 minutes the balloon will be deflated allowing reperfusion and infusion with saline on 4°C will be continued for 10 minutes. After this, a coronary stent will be placed. Primary end points are safety and feasibility of this method.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for this study when they are admitted for acute ST elevation myocardial infarction with a total ST-segment deviation of more than 5 mm and presenting within 6 hours after onset of complaints.

Patients should have a TIMI 0, 1 or 2 flow in the infarction related artery.

Exclusion Criteria:• Age < 18 year

* Cardiogenic shock or pre-shock
* Poor clinical condition with concomitant inconvenience like repeated vomiting, severe chest pain or elsewise according to the judgment of the treating interventionalist.
* Patients with previous myocardial infarction in the culprit area of with previous bypass surgery
* Tortuous coronary arteries
* Complex or long-lasting primary PCI expected
* Inability to understand and give informed consent either in first instance on the table or in second instance on the coronary care unit.
* Other known myocardial diseases, such as moderate or severe left ventricular hypertrophy or cardiomyopathy
* Pregnancy
* First degree AV-block, Mobitz I and Mobitz II block, trifascicular block, or total AV block, Left- and Right Bundle Branch Block
* Patients in whom no access to the coronary circulation can be obtained by the femoral artery or in whom femoral access was problematic Severe concomitant disease or conditions with a life expectancy of less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
arrhythmia or AV-block (1st, 2nd or 3rd degree) | 0 - 20 minutes
  - Is there a higher incidence of rhythm- or conductance disturbances compared with the routine PCI procedure for myocardial infarction or is any other unforeseen side effect observed.
Prolonging of door-to-balloon tome measured in minutes | 30 - 60 minutes
  * Is the protocol easy to perform
  * Is a quick temperature drop achieved (< 5min.) As mentioned earlier, one of the hypotheses for the failure to prove benefit of induced hypothermia in earlier trials, was the relatively long time to achieve the target temperature or the failure to achieve the target temperature at all. Therefore, in this study a quick temperature drop should be recorded in the temperature wire placed distal to the coronary occlusion. A quick temperature drop is defined as a significant drop in distal coronary temperature (<5 °C) within 5 minutes after start of the infusion.
  * After reaching the targeted temperature, is it possible to obtain a stable coronary temperature during 20 minutes.
  * How long is he Door-to-balloon time delayed

SECONDARY OUTCOMES:
Time to target temperature in seconds | 0 - 20
  Time to target temperature

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
by publishing the results in a peer reviewed journal

REFERENCES:
- [Background] Tissier R, Ghaleh B, Cohen MV, Downey JM, Berdeaux A. Myocardial protection with mild hypothermia. Cardiovasc Res. 2012 May 1;94(2):217-25. doi: 10.1093/cvr/cvr315. Epub 2011 Nov 29. PMID 22131353
- [Background] Otterspoor LC, Van't Veer M, van Nunen LX, Wijnbergen I, Tonino PA, Pijls NH. Safety and feasibility of local myocardial hypothermia. Catheter Cardiovasc Interv. 2016 Apr;87(5):877-83. doi: 10.1002/ccd.26139. Epub 2015 Aug 13. PMID 26269225